CLINICAL TRIAL: NCT01979887
Title: Characterization of Signs and Symptoms of Participants With and Without Meibomian Gland Dysfunction
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 195263-007
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Meibomian Glands

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tears
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-MGD Participants: Participants without MGD who have meibum expressed as per protocol. No investigational drug is administered in this study.
  Interventions: Procedure: Meibum Expression
- Mild-Moderate MGD Participants: Participants with Mild-Moderate MGD who have meibum expressed as per protocol. No investigational drug is administered in this study.
  Interventions: Procedure: Meibum Expression
- Severe MGD Participants: Participants with Severe MGD who have meibum expressed as per protocol. No investigational drug is administered in this study.
  Interventions: Procedure: Meibum Expression

INTERVENTIONS:
Procedure: Meibum Expression — Meibum expression as per protocol. No investigational drug is administered in this study.

SUMMARY:
This is an exploratory study to evaluate endpoints used to characterize participants with and without meibomian gland dysfunction (MGD) and will evaluate the correlation between signs and symptoms of MGD. No investigational drug will be administered in this study.

ELIGIBILITY:
Inclusion Criteria:

-Participants characterized as with or without Meibomian Gland Dysfunction.

Exclusion Criteria:

* Lid heating therapy, therapeutic gland expression, or meibomian gland probing within 12 months of enrollment
* Contact lens use in the 30 days prior to enrollment
* Lid hygiene within 48 hours prior to enrollment
* Use of eye makeup within 8 hours of enrollment
* Eyelash growth-stimulating products within 30 days prior to enrollment
* Use of systemic vitamins and/or systemic supplements containing omega 3 fatty acids within 60 days of enrollment
* Use of systemic anti-histamines within 30 days prior to enrollment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants characterized as with or without Meibomian Gland Dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Meibum Quality Score in the Study Eye as Assessed by the Investigator Using a 4-Point Scale | Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Houston, Texas, United States
- London, United Kingdom

REFERENCES:
- [Derived] Ajouz L, Hallak J, Naik R, Nguyen A, Zhao C, Robinson MR, Nichols KK. Evaluation of the Impact of Meibomian Gland Dysfunction Using a Novel Patient-Reported Outcome Instrument. J Ocul Pharmacol Ther. 2024 Jan-Feb;40(1):48-56. doi: 10.1089/jop.2023.0080. Epub 2023 Nov 1. PMID 37910805
- [Derived] Ajouz L, Nguyen A, Zhao C, Robinson MR, Nichols KK. Exploring Signs and Symptoms Associated with Meibomian Gland Dysfunction for Use as Clinical Trial Endpoints. J Ocul Pharmacol Ther. 2023 Nov;39(9):611-621. doi: 10.1089/jop.2023.0064. Epub 2023 Aug 29. PMID 37643299
- [Derived] Nagar S, Ajouz L, Nichols KK, Kumar S, Zhao C, Naidoo KK, Robinson MR, Borchman D. Relationship Between Human Meibum Lipid Composition and the Severity of Meibomian Gland Dysfunction: A Spectroscopic Analysis. Invest Ophthalmol Vis Sci. 2023 Jul 3;64(10):22. doi: 10.1167/iovs.64.10.22. PMID 37466951